CLINICAL TRIAL: NCT00873028
Title: Inspiratory Muscle Strength as a Determinant of Functional Capacity Early After Coronary Artery Bypass Graft Surgery
Brief Title: Evaluation of Inspiratory Muscle Strength Early After Coronary Artery Bypass
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Ricardo Stein, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P1CRh
Record Dates: First submitted 2009-03-30; First posted 2009-04-01 (Estimated); Last update posted 2009-04-01 (Estimated); Status verified 2009-03

CONDITIONS: Coronary Artery Disease
Keywords: Physical therapy; Inspiratory muscles; Exercise
MeSH Terms: conditions — Coronary Artery Disease; Motor Activity | interventions — Cardiac Rehabilitation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Other: In Hospital Cardiopulmonary Rehabilitation
- 2 (No Intervention): Those patients assigned to Control were followed by their own physicians, received routine nursing assistance, were visited daily by the one of the investigators (CPM), but were not exposed to any specific respiratory or motor physical intervention.

INTERVENTIONS:
Other: In Hospital Cardiopulmonary Rehabilitation — The program consisted of bronchial hygiene characterized by detachment and removal of secretions and respiratory exercises which were applied in the respiratory muscles in order to strengthen and increase the resistance. Patients were instructed to maintain diaphragmatic breathing, at a rate of 12 to 18 breaths per minute during EPAP mask use, and the expiratory pressure was increased progressively in the following fashion: 3-8 cm H2O during 3-12 minutes. Also, they performed flexion/extension of hip and knee, active free exercises for upper limbs, ambulation exercise and ascent/descend of stairs
  Other Names: Cardiac rehabilitation; Phase one cardiac rehabilitation
  Arms: 1

SUMMARY:
The purpose of this study is to evaluate the effects of a 6-day postoperative in hospital cardiopulmonary rehabilitation program on inspiratory muscle strength and its potential association with improved functional capacity after coronary artery bypass grafting surgery.

DETAILED DESCRIPTION:
Eligible patients were randomized to a cardiopulmonary rehabilitation program (Rehab; n = 10) or to usual care (Control; n = 10). The randomization was done by the Graphpad StatMate computerized program. Those patients assigned to Control were followed by their own physicians, received routine nursing assistance, were visited daily by the one of the investigators (CPM), but were not exposed to any specific respiratory or motor physical intervention. Those randomized to Rehab received the same medical and nursing care, but followed a structured physical therapy program twice a day.

ELIGIBILITY:
Inclusion Criteria:

* Previous history of more than one vessel coronary artery disease
* Lifelong abstinence from tobacco
* Formal indication for CABG

Exclusion Criteria:

* Patients older than 75 years of age
* Chronic renal failure (dialysis for more than 3 months)
* Unstable angina in the 48 hours prior to CABG
* Moderate or severe valve disease
* Complex cardiac arrhythmia's
* Stroke
* Inability to exercise the lower limbs
* Previous pulmonary disease (forced vital capacity [FVC] < 80% of predicted and/or forced expiratory volume in 1 s [FEV1] < 70% of predicted)
* Previous history of asthma.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-08; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Maximal inspiratory and expiratory pressure were measured (before, 7 and 30 days after surgery). | From 1 day before surgery up to 30 days after surgery (CABG)

SECONDARY OUTCOMES:
Six-minute walk test (6MWT) was performed 7 days after surgery, and maximal cardiopulmonary exercise testing (CPET) was performed 30 days after CABG. | From 7 days after surgery up to 30 days after surgery (CABG)

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Stein, MD.ScD., Principal Investigator — Hospital de Clinicas de Porto Alegre
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Result] Haeffener MP, Ferreira GM, Barreto SS, Arena R, Dall'Ago P. Incentive spirometry with expiratory positive airway pressure reduces pulmonary complications, improves pulmonary function and 6-minute walk distance in patients undergoing coronary artery bypass graft surgery. Am Heart J. 2008 Nov;156(5):900.e1-900.e8. doi: 10.1016/j.ahj.2008.08.006. Epub 2008 Oct 5. PMID 19061704
- [Result] Hirschhorn AD, Richards D, Mungovan SF, Morris NR, Adams L. Supervised moderate intensity exercise improves distance walked at hospital discharge following coronary artery bypass graft surgery--a randomised controlled trial. Heart Lung Circ. 2008 Apr;17(2):129-38. doi: 10.1016/j.hlc.2007.09.004. Epub 2007 Dec 3. PMID 18060837
- [Result] Dall'Ago P, Chiappa GR, Guths H, Stein R, Ribeiro JP. Inspiratory muscle training in patients with heart failure and inspiratory muscle weakness: a randomized trial. J Am Coll Cardiol. 2006 Feb 21;47(4):757-63. doi: 10.1016/j.jacc.2005.09.052. Epub 2006 Jan 26. PMID 16487841
- [Result] Borghi-Silva A, Mendes RG, Costa Fde S, Di Lorenzo VA, Oliveira CR, Luzzi S. The influences of positive end expiratory pressure (PEEP) associated with physiotherapy intervention in phase I cardiac rehabilitation. Clinics (Sao Paulo). 2005 Dec;60(6):465-72. doi: 10.1590/s1807-59322005000600007. Epub 2005 Dec 12. PMID 16358136
- [Result] Herdy AH, Marcchi PL, Vila A, Tavares C, Collaco J, Niebauer J, Ribeiro JP. Pre- and postoperative cardiopulmonary rehabilitation in hospitalized patients undergoing coronary artery bypass surgery: a randomized controlled trial. Am J Phys Med Rehabil. 2008 Sep;87(9):714-9. doi: 10.1097/PHM.0b013e3181839152. PMID 18716482